CLINICAL TRIAL: NCT02533362
Title: A Phase 2, Open-Label, Single Center, Efficacy, Safety, Tolerability, and Pharmacokinetic Study of ANF-Rho™ in Patients With Chronic Neutropenia
Brief Title: ANF-Rho in the Treatment of Chronic Neutropenia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prolong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGCN-002
Record Dates: First submitted 2015-08-10; First posted 2015-08-26 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2015-08

CONDITIONS: Neutropenia, Severe Chronic
MeSH Terms: conditions — Neutropenia, severe chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ANF-Rho (Experimental): pegfilgrastim Anti-Neutropenic Factor (ANF)
  Interventions: Drug: ANF-Rho

INTERVENTIONS:
Drug: ANF-Rho — Pegylated version of recombinant human granulocyte-colony stimulating factor (G-CSF)
  Other Names: pegfilgrastim ANF

SUMMARY:
A 6 month safety, tolerability, efficacy and pharmacokinetic study with ANF-Rho to treat patients with chronic neutropenia.

DETAILED DESCRIPTION:
Chronic neutropenia patients who are eligible for participation will be screened and enrolled to received open-label ANF-Rho for a period of 6 months. Study participation will be separated into 2 periods, Induction (8 weeks) and Maintenance (16 weeks). Blood samples to measure neutrophil levels and biochemistry labs will be drawn throughout the study to monitor efficacy response and patient safety. Pharmacokinetic samples will be collected during both periods and questionnaires will be completed by the patient and investigator for bone pain, quality of life (QOL) and injection site reaction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 1 years of age or older
2. Patients with established chronic neutropenia defined as Median Absolute Neutrophil Count (ANC) < 0.5 x 109/L (both with and without demonstrated genetic lesion) having an indication for treatment, including:

   Independent of hematological parameters, all patients with: Shwachman-Diamond syndrome (SDS), Barth's syndrome or other inherited diseases associated with neutropenia (exclude Glycogen Storage Disease 1b)
3. Patients on granulocyte-colony stimulating factor (GCSF) & PEG-GCSF treatment are still eligible to participate after a washout period of 7 days, after the stopping of the drug
4. Signed and dated informed written consent/assent by the patient/parent
5. Women of childbearing potential with a negative serum pregnancy test and using a reliable method of contraception during the study period. Male study participants also agreeing to use contraception for the study period.

Exclusion Criteria:

1. Evidence of chromosomal abnormalities, myelodysplasia, hematologic malignancy, aplastic anemia, systemic lupus erythematosus, or rheumatoid arthritis (Felty's syndrome) or if the neutropenia was drug-induced
2. Progressive malignant disease or malignancy history
3. Presence of macrophage activation syndrome before the diagnosis of neutropenia
4. Clinical Significant Abnormal Renal, Cardiac, Hepatic or Blood Coagulation disease.
5. Chronic infection such as hepatitis B virus (HBV), hepatitis C Virus (HCV) or Human immunodeficiency virus( HIV) or history of tuberculosis
6. Association with anemia, thrombocytopenia (low blood platelets) before the diagnosis of neutropenia.
7. Drug abuse, substance abuse, or alcohol abuse
8. Use of any other investigational drug at the time of enrollment, or within 5 half-lives prior to enrollment, whichever is longer
9. Patients unwilling and/or who are not capable of ensuring compliance with the provisions of the study protocol
10. Women who are pregnant or breastfeeding
11. Women of childbearing potential who do not use an approved method of birth control. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods) is not acceptable
12. Patients with known DNA loss-of-function mutations in GCSFR and RUNX1 genes

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Neutrophil response rate to ANF Rho following a 6 month treatment period (induction, stabilization and maintenance periods) in patients with Chronic Neutropenia. | 6 months
  Median Absolute Neutrophil Count (ANC) of ≥1.0 x 109/L over the 6 months total treatment period

SECONDARY OUTCOMES:
Serum concentration of ANF-Rho over time | 6 months
  Pharmacokinetic parameter measuring ANF-Rho levels over time
The peak plasma concentration of ANF-Rho after administration (Cmax) over time | 6 months
  Pharmacokinetic Parameter measuring ANF-Rho levels over time
Total ANF-Rho exposure (AUC) | 6 months
  Pharmacokinetic parameter measuring ANF-Rho levels from time 0 through last dose.
Time to peak plasma concentration of ANF-Rho (Tmax) | 6 months
  Pharmacokinetic parameter measuring the time to Cmax.
Half-Life of ANF-Rho (T1/2) | 6 months
  Pharmacokinetic parameter to measure the time required for the concentration of the drug to reach half of its original value
Rate of subject reported infection related morbidities (infections, hospitalisations and antibiotic use) in Chronic Neutropenia patients treated with ANF Rho | 6 months
Evaluate the effect of ANF Rho on the Quality of Life and Bone Pain in Chronic Neutropenia patients. | 6 months
  Change in Quality of life over 6 months measured by the Short Form 36, change in bone pain over 6 months measured by the Bone Pain Questionnaire, Wong and Baker Scale and FLACC Behavioral Pain Assessment Scale
Evaluate safety and tolerability of subcutaneous injections of ANF Rho in chronic neutropenia patients. | 6 months
  Composite endpoint with multiple vital signs, bone scans, biopsies, splenic ultrasounds, electrocardiographic assessments, clinical signs, and bio-analytical measures (e.g., biochemistry), and reported adverse events following repeated dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Hemant Misra, PhD, Study Director — Prolong Pharmaceuticals